CLINICAL TRIAL: NCT07052513
Title: Modified Autologous Leukocyte Cells for the Treatment of Acute Kidney Injury After Cardiac Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M2RLAB SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2R.AKI.2021; 2023-504610-30-01 (EU CTIS Number)
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Acute Kidney Injury
Keywords: Cardiac Surgery; Thoracic Surgery; Acute Renal Insufficiency; Acute Renal Injury; Major Adverse Kidney Event; Autologous Leukocyte Cells; Leukocyte Cells; Autologous Mononuclear Cells; Mononuclear Cells; Acute Kidney Disease
MeSH Terms: conditions — Acute Kidney Injury | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be assigned to one of the two treatment groups in a 1:1 ratio. In both groups an intravenous injection will be administered to maintain the blinding of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline Solution for injection (Placebo Comparator): Participants randomized to placebo will receive a single 10 mL dose Intravenous (IV) infusion of normal saline (0.9 percent) no later than 36 hours after the participant's diagnosis of AKI and inclusion in the study.
  Interventions: Drug: Placebo
- Cell therapy with leukocyte cells from the participant himself/herself (Experimental): Participants randomized to experimental group will receive a single 10 mL dose IV of leukocyte cells concentration of 6-15.4 x10^6 cells/mL no later than 36 hours after the participant's diagnosis of AKI and inclusion in the study.
  Interventions: Drug: M2RLAB 001

INTERVENTIONS:
Drug: Placebo — Intravenous infusion of normal saline.
  Other Names: Saline Solution
  Arms: Saline Solution for injection
Drug: M2RLAB 001 — Intravenous infusion of M2RLAB 001
  Other Names: Autologous Leukocyte Cells
  Arms: Cell therapy with leukocyte cells from the participant himself/herself

SUMMARY:
The purpose of this clinical trial is to assess the efficacy and safety of cell therapy with modified leukocyte cells from the participant himself/herself versus placebo in patients who develop Acute Kidney Injury (AKI) within the first 48 hours after cardiac surgery.

The main questions it aims to answer are:

* Does cell therapy reduce the recovery time of kidney function?
* What medical problems do participants have when receiving cell therapy?

Researchers will compare cell therapy with a placebo (a look-alike substance that contains no drug) to see if cell therapy works to treat AKI. The safety of cell therapy with leukocyte cells will also be studied.

DETAILED DESCRIPTION:
This is a Phase II, multi-center, randomized, placebo-controlled clinical trial, with 2 treatment arms and single blind. After being informed about the study, participants who meet the eligibility criteria will be randomized in 1:1 ratio to treatment with a single administration of cell therapy with leukocyte cells from the participant himself/herself or placebo (approximately 49 subjects per group).

Acute kidney injury (AKI) is one of the main complications after cardiac surgery. In fact, AKI after cardiac surgery is associated with high morbidity and mortality. Currently, there are no effective therapies for kidney injury after cardiac surgery, but there is evidence that recovery is possible if the injury processes are overcome. Thus, due to the lack of preventive and therapeutic options at present, cell therapy has gained importance in recent years in different clinical trials. Thus, within this context, the use of modified leukocyte cells as cell therapy is also an alternative for the treatment of AKI due to their powerful immunomodulatory effect. On the other hand, the use of placebo is justified because there is currently no other pharmacological treatment available to serve as an active control. A placebo-controlled study is optimal to evaluate the efficacy and safety of an experimental treatment.

Researchers hypothesized that cell therapy with autologous leukocyte cells can be safe, well tolerated and clinically beneficial versus placebo for participants who develop AKI within the first 48 hours after cardiac surgery.

This study consists of 3 phases: the initial phase, the observation phase, and the follow-up phase. The total duration of each participant in the trial will be 3 months:

* Initial phase: The patient undergoing cardiac surgery will sign the informed consent (IC) before the surgery (at a scheduled visit prior to his/her hospitalization or at the time of his/her hospitalization and prior to undergoing the procedure). As indicated in the Inclusion criteria, only participants who present AKI within the first 48 hours post cardiac surgery will be included. The participants who meet all the inclusion criteria and none of the exclusion criteria will be randomized in a 1:1 ratio to one of the two study groups. A volume of at least 60 mL of peripheral blood will be extracted from the patient, from which the cell therapy will be prepared (in cases where the patient is included in the experimental group) The investigational product/placebo will be administered to the patient within 36 hours of AKI diagnosis.
* Observation phase: It includes the period from when the patient receives the investigational drug/placebo until he or she is discharged from the hospital. This period lasts 16 to 20 days, depending on the clinical evolution of the participants. During this phase, participants will be followed and will undergo different tests in order to evaluate the effectiveness and safety of the investigational treatment vs. placebo.
* Follow-up phase: It includes the period from when the patient receives hospital discharge and ends 90 days from the date of inclusion of the participant in the study. At this stage, participants will be monitored to evaluate the efficacy and safety of the experimental cell therapy drug vs. placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants older than 18 years of age, being able to understand and sign the Informed Consent.
2. Participants undergoing elective valvular and/or coronary cardiac surgery performed with extracorporeal circulation.
3. Present pre-operative AKI risk more or equal to 30 percent according to the Leicester Cardiosurgery scale.
4. Present AKI within the first 48 hours post cardiac surgery in one of the following classifications defined by the AKIN scale (Acute Kidney Injury Network):

   AKIN 1: An increase in serum creatinine by at least 0.3 mg/dL (more or equal to 26.4 micromol/L) from baseline, or an increase to more or equal to 150-200 percent (corresponding to a 1.5- to 2-fold increase) from baseline. In addition, the patient must have a positive acute tubular necrosis score within the first 48 hours post cardiac surgery, defined as the presence of at least 3 of the following 4 scenarios: Sodium excretion fraction more than 2 percent, urinary osmolality lower than 400 mOsm/kg, urine sodium more than 40 mmol/L, presence of shock or nephrotoxic agents.

   AKIN 2: An increase in serum creatinine to more than 200 percent and up to a maximum of 300 percent (corresponding to an increase of more than 2 and up to 3 times) over baseline.

   AKIN 3: An increase in serum creatinine to more than 300 percent (corresponding to more than 3-fold increase) over baseline, or an increase in serum creatinine levels to more or equal to 4.0 mg/dl (more or equal to 354 micromol/l) with an acute increase of at least 0.5 mg/dl (44 micromol/l).
5. In the case of women or men of childbearing age, for safety, those who undertake to follow the contraceptive measures required from their discharge from hospital until the end of their participation in the clinical trial.

Exclusion Criteria:

1. Chronic Kidney Disease (CKD) in stage IV or V (glomerular filtration rate [GFR] less than 30 ml/min).
2. AKI one month prior to heart surgery.
3. Participants who have previously undergone renal therapy.
4. Participants who are scheduled to start renal replacement therapy within the next 72 hours.
5. Interstitial glomerulonephritis or vasculitis.
6. Pregnancy.
7. Women in breastfeeding period
8. Renal transplant history.
9. Endocarditis.
10. Participants with mechanical assistance devices: extracorporeal membrane oxygenation (ECMO), left ventricular assist device (LVAD), right ventricular assist device (RVAD), intra-aortic balloon pumps (IABP).
11. Known severe ventricular dysfunction (left ventricular ejection fraction [LVEF] less than 30 percent).
12. Post-surgical septic infectious condition.
13. Positive serology for hepatitis C virus (HCV), hepatitis B virus antigen (HBSAg), human immunodeficiency virus (HIV) or syphilis (by VDRL/TP: Venereal Disease Research Laboratory/Treponema pallidum). This criterion will be assessed once it has been confirmed that the patient has developed AKI.
14. Participants enrolled in another clinical trial testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-07-17 (Estimated); Primary Completion 2027-06-17 (Estimated); Study Completion 2027-09-02 (Estimated)

PRIMARY OUTCOMES:
Recovery time of kidney function | Baseline Phase (Day 0), Observation Phase: From Visit 1 (1 day after treatment) to Visit 7 (7 days after treatment)
  Time (in days) to recovery of the creatinine to baseline values (in the range of more or less than 30 percent from baseline).
Proportion of participants with persistently altered creatinine values (more than 31 percent from baseline values) 7 days after AKI episode | Baseline Phase (Day 0), Observation Phase: From Visit 1 (1 day after treatment) to Visit 7 (7 days after treatment
  Measured as the incidence of Acute Kidney Disease (AKD): persistence of altered creatinine values 7 days after the AKI episode.
Occurrence of adverse events (AEs) | Up to Day 90
  Number of AEs reported.
Occurrence of serious AEs (SAEs) | Up to Day 90
  Number of SAEs reported
Occurrence of AEs resulting in discontinuation of study treatment | Up to Day 90
  Number of AEs resulting in discontinuation of study treatment reported
Occurrence of AEs of special interest (AESIs) | Up to Day 90
  Number of AESIs reported.

SECONDARY OUTCOMES:
Major Adverse Kidney Events (MAKE) incidence reduction | Baseline Phase: Day 0, Observation Phase: From Visit 1 (1 day after treatment) to Visit 7 (7 days after treatment) and Follow-up phase: Day 30 and 90
  Proportion of patients with MAKE incidence reduction. MAKE is considered as the development of events related to disease progression, which is defined as death related to renal failure, need for dialysis or permanent reduction of estimated Glomerular Filtration Rate more than 30 percent since baseline
Time to appear of Major Adverse Kidney Events (MAKE) | Up to Day 90
  Time to appear of MAKE. MAKE is considered as the development of events related to disease progression, which is defined as death related to renal failure, need for dialysis or permanent reduction of estimated Glomerular Filtration Rate more than 30 percent since baseline
Number of participants on renal replacement therapy | Up to Day 90
  Number of participants requiring dialysis
Renal replacement therapy duration. | Up to Day 90
  Time (in days) of the required dialysis.
Duration of admission to Intensive Care Unit (ICU) | Up to Day 90
  Time (in days) of ICU stay of participants.
Duration of hospital stay | Up to Day 90
  Time (in days) of hospital stay of participants.
Patient survival after 30 days | Up to Day 30
  Proportion of participants who survived after 30 days.
Patient survival after 90 days | Up to Day 90
  Proportion of participants who survived after 90 days.
Participants requiring dialysis versus participants who survived without requiring dialysis after 30 days | Up to Day 30
  Proportion of participants who survived requiring dialysis versus participants who survived without requiring dialysis after 30 days post cardiac surgery.
Participants requiring dialysis versus participants who survived without requiring dialysis after 90 days | Up to Day 90
  Proportion of participants who survived requiring dialysis versus participants who survived without requiring dialysis after 90 days post cardiac surgery.
Maximum creatinine values (peak creatinine) recorded during participants' hospitalization | Baseline Phase: Day 0 and Observation Phase: From Visit 1 (1 day after treatment) to Visit 7 (7 days after treatment)
  Maximum creatinine value (peak creatinine) recorded. Creatinine levels will be measured in serum.
Time (day) of maximum creatinine values (peak creatinine) recorded during participants' hospitalization | Baseline Phase: Day 0 and Observation Phase: From Visit 1 (1 day after treatment) to Visit 7 (7 days after treatment)
  Day of maximum creatinine values (peak creatinine) recorded. Creatinine levels will be measured in serum.
Improvement in levels of injury biomarkers in urine | Baseline Phase: Day 0 and Observation Phase: Visit 7 (7 days after treatment)
  Proportion of participants with variations of more than 30 percent in the values of injury biomarkers in urine [Albumin and Neutrophil gelatinase-associated lipocalin (NGAL)]
Participants presenting surgical wound infections | Up to Day 90
  Proportion of participants with surgical wound infections.
Participants presenting respiratory infections during ICU stay | Up to Day 90
  Proportion of participants with respiratory infections during ICU stay.
Participants who present complications related to surgery | Up to Day 90
  Proportion of participants with any complication related to surgery (Sternotomy, Reintervention, Circulatory support).
Number of complications related to surgery | Up to Day 90
  Absolute number of any complication related to surgery (Sternotomy, Reintervention, Circulatory support).
Unexplained haemodynamic worsening | Observational Phase: Day 1 and Day 7
  Unexplained haemodynamic worsening measured as: drop in cardiac index to less than 2.5 L/min/m^2 (if it was previously higher), drop in systemic systolic blood pressure more than 30 percent or to less than 90 mmgHg, and/or more than 30 increase in vasoactive drugs dose.

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Poch López de Briñas, Principal Investigator — Hospital Clinic of Barcelona; Francisco José Roca Oporto, Principal Investigator — Hospital Univ. Virgen del Rocío
Locations (2):
- Spain (2):
  - Hospital Univ. Virgen del Rocío, Seville, Andalusia
  - Hospital Clinic of Barcelona, Barcelona, Catalonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jativa S, Torrico S, Calle P, Munoz A, Garcia M, Larque AB, Poch E, Hotter G. NGAL release from peripheral blood mononuclear cells protects against acute kidney injury and prevents AKI induced fibrosis. Biomed Pharmacother. 2022 Sep;153:113415. doi: 10.1016/j.biopha.2022.113415. Epub 2022 Jul 18. PMID 36076483
- [Background] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245